CLINICAL TRIAL: NCT06774079
Title: A Randomized Clinical Trial to Determine the Effect of Dual Glucose-dependent Insulinotropic Polypeptide (GIP)/GLP-1 Receptor Agonist-mediated Weight Loss and Diet on Crohn's Disease Clinical Response: a Pilot Study
Brief Title: Glucagon-like Peptide-1 Receptor Agonist (GLP-1 RA) and Diet in Inflammatory Bowel Disease (IBD) Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Oriana Mazorra Damas, Associate Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20240982
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
Keywords: inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Tirzepatide; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide group (Experimental): Participants will be in this group for up to 12 weeks.
  Interventions: Drug: Tirzepatide; Behavioral: Mediterranean diet
- Mediterranean diet group (Experimental): Participants will be in this group for up to 12 weeks.
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Drug: Tirzepatide — Patients in this arm will receive tirzepatide starting at 2.5 mg subcutaneous (SC) weekly for 4 weeks, then increase to 5 mg SC weekly for 4 weeks and then 7.5 mg SC weekly for the last 4 weeks of the intervention period. Place of injection includes abdomen, thigh, or upper arm.
  Arms: Tirzepatide group
Behavioral: Mediterranean diet — The diet is comprised of a content of 25-30 grams of fiber per day (from fruits, vegetables, whole grains) that is low in animal protein and minimally processing of foods The diet arm will receive dietary guidance from our dietician on weekly 30-minute guided sessions. Participants will be encouraged to adhere to the diet for up to three meals per day for the duration of the study.

SUMMARY:
The purpose of this study is to use diet and an injectable medication called tirzepatide (Zepbound) glucose-dependent insulinotropic polypeptide and glucagon-like peptide-1 receptor agonist (GIP-GLP-1 RA) medication as adjunctive therapy (another treatment used together with the primary treatment) for Crohn's disease patients with mild disease who are on stable doses of biologic medication (infliximab or adalimumab) and who have a body mass index (BMI) of at least 27.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Confirmed diagnosis of Crohn's disease
* Mildly active disease, defined by clinical symptoms using the Harvey Bradshaw Index (HBI) score between 5 and 7 (the HBI is a continuous score ranging from 0-16 where <4 is considered remission)
* BMI ≥ 27 kg/m2
* Patients will be on stable doses of medical therapy (anti-tumor necrosis factor (TNF) alpha blockers)

Exclusion Criteria:

* Patients under 18 years of age
* Patients with ulcerative colitis
* Patients with infectious colitis
* BMI<27 kg/m2
* Patients with type 1 or type 2 diabetes
* Contraindications to a GIP/GLP-1 RA, including patients with a personal or family history of medullary thyroid cancer or in patients with Multiple Endocrine Neoplasia syndrome type 2
* Patients already on GIP/GLP-1 RA therapy
* Patients with the following chronic symptoms: severe constipation, nausea, and/or vomiting
* Patients with the following medical history: small bowel obstruction in the last year, intestinal stricture, known or suspected diagnosis of gastroparesis
* Adults unable to consent
* Pregnant patients (will be confirmed via a pregnancy test)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of participants retained | Baseline, 12 weeks
  The percentage of participants retained will be measured
Number of patients who adhere to diet measured by 24 hour dietary recall | Up to 12 weeks
  Number of patients who adhere to diet measured by 24 hour dietary recall
Number of patients who adhere to medications measured by self report | Up to 12 weeks
  Number of patients who adhere to medications measured by self report

SECONDARY OUTCOMES:
Number of calls completed | Up to 12 weeks
  Number of calls completed. Calls will be made either on a phone or virtually using Zoom.
Number of dietary recall (ASA24) surveys completed | Up to 12 weeks
  Number of dietary recall (ASA24) surveys completed
Number of clinical symptom (HBI/CDAI) surveys completed | Up to 12 weeks
  Number of clinical symptom (HBI/CDAI) surveys completed
Number of blood samples completed | Up to 12 weeks
  Number of blood samples completed
Number of stool samples completed | Up to 12 weeks
  Number of stool samples completed

CONTACTS AND LOCATIONS:
Overall Officials: Oriana Damas, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No